CLINICAL TRIAL: NCT04044963
Title: The Effect of a Prehabilitation Exercise Program on Physical Functioning for Patients Undergoing Kidney Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Nguan, Associate Professor - UBC Department of Urologic Sciences. Program Director - UBC Urology Postgraduate Education. Surgical Director - Kidney Transplant Program, Vancouver General Hospital, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H19-01405
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: End Stage Renal Disease
Keywords: Renal transplantation; Prehabilitation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Exercise; Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): All participants who are allocated to the exercise group will be asked to complete 4-5 days per week of mixed modality exercise incorporating aerobic, resistance, and flexibility training. The exercise intervention is prescribed based on the FITT principle: frequency, intensity, time and type. The 10-point Rating of Perceived Exertion (RPE) scale, which has been well correlated to target HR levels, will be used to monitor exercise intensity levels throughout the intervention, with participants instructed to maintain their intensity level at 3-5 during exercise sessions. Participant progression will be individualized and based on their subjective perceived intensity level using the RPE scale. In person instruction, from a member of the research team with standard first aid and CPR-C training, and an instructional handout and exercise log will be provided, as well as exercise resistance bands to perform resistance exercises.
  Interventions: Behavioral: Exercise and Prehabilitation
- Control Group (No Intervention): This will consist of regular care, which is standard procedure.

INTERVENTIONS:
Behavioral: Exercise and Prehabilitation — All participants who are allocated to the exercise group will be asked to complete 4-5 days per week of mixed modality exercise incorporating aerobic, resistance, and flexibility training. The aerobic component can include any modality the patient is capable of doing, including walking, swimming or biking. By the end of the prehabilitation period the target will be 30 minutes of aerobic exercise three times a week at an intensity of 3-5 RPE. The resistance component will include 5-6 exercises using body weight and resistance bands. The target will be 12 repetitions and 3 sets, two times a week. The flexibility component will include 5 exercises that can be completed at the end of each session.
  Participants will self-report their participation in the prehabilitation program based on an electronic survey.
  Arms: Exercise Group

SUMMARY:
Pre-operative physical functioning has been acknowledged as a factor influencing post-operative complication risk, recovery progression and mortality risk. Current guidelines have yet to focus on the pre-operative period as a potential target to improve levels of physical functioning before renal transplantation. This project proposes the introduction of an exercise intervention pre-operatively to mitigate functional decline pre-operatively and improve post-operative outcomes following renal transplantation.

We hypothesize that a home-based exercise prehabilitation program prior to kidney transplantation will result in improved functional outcomes including the 6-minute walk test, 60-second timed sit to stand, Fried Frailty Score, quality of life and fatigue. Further we hypothesize that prehabilitation will result in improved outcomes regarding post-operative recovery, complication rate, length of stay and mortality.

Objectives

A) Identify whether a prehabilitation program can mitigate functional decline pre-operatively regarding walking speed, strength, endurance, quality of life and fatigue

B) To determine whether a tailored home-based exercise program prior to kidney transplantation is feasible with regards to adherence in patients with Chronic Kidney Disease (CKD) and End Stage Renal Disease (ESRD).

C) To determine if a prehabilitation program results in improved clinical outcomes within one week following Kidney Transplantation (KT) as well as at 30 and 90 days including but not limited to time to first ambulation, time to first bowel movement, postoperative complications (Clavien-Dindo classification), mortality and length of stay.

D) Quantify the differences described above, if any exist.

DETAILED DESCRIPTION:
This is a pilot study involving kidney transplant recipients who will be receiving a kidney from a live donor and receiving care at Vancouver General Hospital or St. Paul's Hospital.

Upon enrollment baseline demographics, including age, sex, BMI, ethnicity will be recorded. Baseline physical measures will include resting HR and BP, 6-minute walk test (6-MWT) (measuring HR and RPE every minute throughout), 30-second timed sit to stand (HR and RPE at the end), Fried Frailty score (Subjective: weight loss, energy level, physical activity levels - Objective: weakness, slowed walking speed), and a quality of life (QOL) and fatigue survey. These baseline measures will be recorded at onset of enrollment, every 3 months, again 1 week prior to KT, 4 weeks post operatively, and each month after for 5 months. This will add up to 6 months of follow up. The patient reported outcomes - post-op recovery survey and fatigue survey will also be completed on day 2 and day 5 post-operatively as well as 1, 2 and 4-weeks post-operatively.

Questionnaire Administration:

All questionnaires will be available electronically using Qualtrics as well via a paper copy. These will be administered based on patient preference; they will both be administered either electronically using Qualtrics or via a paper copy.

Participant Expectations: Assessment and Follow-up

Baseline Assessment:

Physical Fitness assessment (6-MWT, 30-sec sit to stand, Fried Frailty Score, HR+BP), Quality of Life Survey, Fatigue Survey, Baseline Exercise Level Questionnaire

Every 3 Months Leading Up to Renal Transplant:

I.e. 3-month, 6-month, 9-month, 12-month post baseline assessment - Physical Fitness assessment (6-MWT, 30-sec sit to stand, Fried Frailty Score, HR+BP), Quality of Life Survey, Fatigue Survey

One-week Prior to Renal Transplant:

Physical Fitness assessment (6-MWT, 30-sec sit to stand, Fried Frailty Score, HR+BP), Quality of Life Survey, Fatigue Survey

Two Day Post Operation:

Patient Reported Outcomes - Post-op recovery survey

Five Day Post Operation:

Patient Reported Outcomes - Post-op recovery survey

One Week Post Operation:

Patient Reported Outcomes - Post-op recovery survey, Fatigue survey

Two Week Post Operation:

Patient Reported Outcomes - Post-op recovery survey, Fatigue survey

One Month Post Operation:

Patient Reported Outcomes - Post-op recovery survey, Physical Fitness assessment (6-MWT, 30-sec sit to stand, Fried Frailty Score, HR+BP), Quality of Life Survey, Fatigue Survey

Two Month Post Operation:

Physical Fitness assessment (6-MWT, 30-sec sit to stand, Fried Frailty Score, HR+BP)

Three Month Post Operation:

Physical Fitness assessment (6-MWT, 30-sec sit to stand, Fried Frailty Score, HR+BP)

Four Month Post Operation:

Physical Fitness assessment (6-MWT, 30-sec sit to stand, Fried Frailty Score, HR+BP)

Five Month Post Operation:

Physical Fitness assessment (6-MWT, 30-sec sit to stand, Fried Frailty Score, HR+BP)

Six Month Post Operation:

Physical Fitness assessment (6-MWT, 30-sec sit to stand, Fried Frailty Score, HR+BP), Quality of Life Survey, Fatigue Survey

Following the baseline assessment, participants will be randomly allocated to treatment groups (2:1) to a 1) home-based training program (exercise group) and a 2) control group (no prehab just regular care, which is standard procedure). This random allocation will occur via a computer-generated randomized scheme.

Following enrolment, each participant allocated to the exercise group will begin the prehabilitation protocol shortly after the initial consultation with their attending urologist. The prehabilitation protocol will be performed from this initial consult up until the date of the scheduled KT (minimum 4 weeks). In person instruction, from a member of the research team with standard first aid and cardiopulmonary resuscitation (CPR) training, and an instructional handout and exercise log will be provided, as well as exercise resistance bands to perform resistance exercises. The exercise log will be given to each study participant and will be used solely as a method to make organizing and recording each exercise session easier for the participant. The exercise log will not be collected by the study team. The exercise log should be completed following each exercise session and it should take no longer than 2-3 minutes to complete. All participants who are allocated to the exercise group will be asked to complete 4-5 days per week of mixed modality exercise incorporating aerobic, resistance, and flexibility training. The exercise intervention is prescribed based on the FITT principle: frequency, intensity, time and type. The 10-point Rating of Perceived Exertion (RPE) scale, which has been well correlated to target HR levels, will be used to monitor exercise intensity levels throughout the intervention, with participants instructed to maintain their intensity level at 3-5 during exercise sessions. Participant progression will be individualized and based on their subjective perceived intensity level using the RPE scale.

Aerobic Component:

The aerobic component can include any modality the patient is capable of doing, including walking, swimming or biking. By the end of the prehabilitation period the target will be 30 minutes of aerobic exercise three times a week at an intensity of 3-5 RPE. Initially, the patient may start with 10 minutes, three times a week. Slowly progressing first with duration (10 to 15 min), followed by an increase in exercise intensity (increased speed or grade - RPE from 3 - 5).

Resistance Component:

The resistance component will include 5-6 exercises using body weight and resistance bands. The target will be 12 repetitions and 3 sets, two times a week. Initially, the patient may start with 8 repetitions and 1 set and progress to a maximum of 12 repetitions and 3 sets. If a participant is able to complete >12 repetitions and 3 sets of a specific resistance exercise than they will increase resistance (i.e. green band to red band). These exercises will be provided in the handout that each participant will receive. Lower body exercises will include foot, knee and hip flexion and extension, and hip adduction and adduction. Upper body exercises will include arm and wrist flexion and extension, and shoulder abduction and adduction.

Flexibility Component:

The flexibility component will include 5 exercises that can be completed at the end of each session. This should take no longer than 5-10 minutes. These exercises will be provided in the handout that each participant will receive. Flexibility exercises will include a hamstring stretch, quadriceps stretch, hip external rotation, standing lumbar extension, and upper body shoulder and arm stretch.

Participants will self-report their participation in the prehabilitation program based on an electronic survey. The intent of the survey is to follow the frequency, time and type of exercise of the patient leading up to the operation and identify whether the patient is adhering to the exercise intervention. The survey will take an estimated 3-5 minutes to complete and will primarily consist of Likert-scale questions and checkboxes. Survey responses will be stored on University of British Columbia (UBC) owned and operated servers such as the Qualtrics tool supported and maintained by UBC IT.

Self-reported exercise and physical measures will be recorded at baseline, and every two or three weeks prior to each patients KT as well as bi-weekly post-operatively up until 1-month post KT. This confidential, anonymized, electronic pre-operative survey will be used to keep track of self-reported physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to physically participate in a home-based prehabilitation program and all functional outcome measures
2. Ability to read and write in English to respond to study questionnaires
3. Age = to or > 19 and any gender
4. Receiving care at Vancouver General Hospital or St. Paul's Hospital
5. Has been fully worked up for suitability for renal transplantation
6. Received physician clearance to participate

Exclusion Criteria:

1. Unstable pulmonary or symptomatic cardiac disease
2. Recent fracture or acute musculoskeletal injury that precludes the ability to exercise

4. Is unable to understand the purpose of the study, or cannot give written consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk test (6-MWT). | Change from baseline to 1 week prior to renal transplantation. Again, change from 1 month post transplant to 6 month post transplant.
  Change from baseline in metres (m).
Change in 30-second timed sit to stand. | Change from baseline to 1 week prior to renal transplantation. Again, change from 1 month post transplant to 6 month post transplant.
  Change from baseline in number of repetitions completed in 30 seconds.
Change in Fried Frailty Score. | Change from baseline to 1 week prior to renal transplantation. Again, change from 1 month post transplant to 6 month post transplant.
  Change from baseline, score based on a 4-point scale.
Change in fatigue level. | Change from baseline to 1 week prior to renal transplantation. Again, change from 1 month post transplant to 6 month post transplant.
  Change from baseline, score based on a 13 point scale.
Change in quality of life (QOL). | Change from baseline to 1 week prior to renal transplantation. Again, change from 1 month post transplant to 6 month post transplant.
  Change from baseline, score based on a 25 question survey.
Time to first ambulation following kidney transplantation. | One week following kidney transplant.
  Assessed in days.
Time to first bowel movement following kidney transplantation. | One week following kidney transplant.
  Assessed in days.
Change in number of participants with post operative complications. | Change from 1 week following kidney transplant to 30 and 90 days post operatively.
  Number of participants with post operative complications as assessed by Clavien-Dindo classification.
Length of hospital stay following kidney transplantation. | One week following kidney transplant.
  Assessed in days.

SECONDARY OUTCOMES:
Participant adherence to a tailored home-based exercise program. | From date of randomization until the date of kidney transplantation, assessed up to 24 months.
  Exercise tracker questionnaire. Adherence will be calculated based on a 4 point scale assessing frequency, intensity, time and type of exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nguan, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No